CLINICAL TRIAL: NCT05353244
Title: Effects of Personalized Repetitive Transcranial Magnetic Stimulation (PrTMS) on Human Performance and Sleep Quality
Brief Title: Effects of PrTMS on Performance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never commenced.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Victor Finomore, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2111477106
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Sleep Quality; Cognition Improvement
Keywords: PrTMS; EEG; Sleep; Cogniton
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an active or sham intervention group. Each participant will complete 30 PrTMS or sham sessions. Through the course of the 6-week study, participants will be asked to wear a lab-provided sleep tracking ring (Oura).
  Each participant, regardless of group, will complete daily and weekly surveys and assessments including a qEEG and cognitive assessments. At the intake, midpoint, and exit, a battery of surveys will be administered as well.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Principal Investigator, statisticians, and participants will be blinded to the condition (PrTMS vs Sham). Only the providers of the treatment will be aware of the treatment condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active PrTMS (Active Comparator): Participants will receive PrTMS five days a week for six weeks.
  Interventions: Device: PrTMS
- Sham (Sham Comparator): Participants will receive sham treatment five days a week for six weeks.
  Interventions: Device: Sham

INTERVENTIONS:
Device: PrTMS — Each participant will receive a personalized rTMS treatment based on their individual alpha frequency.
  Arms: Active PrTMS
Device: Sham — Using a sham coil that looks and sounds like an actual TMS coil, each participant will receive sham rTMS treatments.
  Arms: Sham

SUMMARY:
The purpose of this study is to assess the ability of a form of non-invasive brain stimulation called personalized repetitive transcranial magnetic stimulation, or PrTMS, to enhance cognitive performance and sleep quality from baseline metrics.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) is an FDA approved, non-invasive, non-pharmaceutical strategy for treating adults with major depression. This particular treatment strategy is also deemed safe and well-tolerated per the numerous clinical trials of over 300 patients. Additionally, the extant literature reports numerous occurrences of human performance enhancement in association with rTMS, such as better visual perception, motor learning, objective identification, attention, memory, as well as faster eye movements. However, recent advancements in rTMS yield promise for a more personalized protocol that is specific to individual needs and is based on quantitative electroencephalography (qEEG), enabling a correlation between qEEG and human behavior, though further investigation is necessary. Therefore, this study will examine personalized qEEG-guided rTMS (PrTMS) based upon each patient's pretreatment qEEG readings.

PrTMS uses neural alpha wave dynamics to target its TMS intervention via PeakLogic software with respect to location and frequency of TMS application. If PrTMS is effective, then researchers should be able to observe specific changes, e.g., more consistent fundamental frequency and increased alpha wave coherence across multiple brain sites, as PrTMS interventions progress. More importantly, alpha wave coherence is known to be associated with improved sleep behavior, cognition, and emotional reactivity. Thus, it is reasonable to hypothesize that changes in neural activity (as detected via qEEG) may result in several positive behavioral and perceptual (e.g., improved mood state/reduced anxiety) responses even for healthy populations.

The goal of PrTMS is to steadily nudge neural alpha wave responses towards a common fundamental frequency (10 to 12 Hz) across all brain regions. These frequencies vary over time, like all natural systems, with larger variations thought to be tied to behavioral symptomologies such as anxiety, PTSD, sleep disturbances and other conditions. Once this goal is achieved, neural activity across the brain is in coherence, which is assumed to be a natural and more efficient state for brain activity, with downstream effects such as the alleviation of symptoms relevant to brain-related disease/injury and/or heightened cognitive function.

Provided the well understood importance of adequate sleep and keen cognition for both the quality of daily living as well as longevity, efforts to thwart any potential disturbances to either offers promise for the betterment of the RNI's targeted populations, AMP2 (Athletics, Military, Patient, and general Population communities). Further, there are very intimate associations between sleep and cognition; put simply, the more one sleeps and the better quality of said sleep, the better one's cognitive skills will be the subsequent day. Indeed, previous research reported improved attentional focus, cognitive processing, and memory development with greater sleep durations. Contrarily, when one is deprived of sleep, one might expect to experience decreased physical performance capabilities (e.g., decreased force production), deleterious effects to glucose metabolism, poor appetite, diminished protein synthesis at the cellular level, as well as increased systemic inflammation. One intriguing strategy for improving sleep and cognition that is both noninvasive and non-pharmaceutical is Transcranial Magnetic Stimulation (TMS). Previous literature suggests that Transcranial Magnetic Stimulation was effective in enhancing both sleep and cognitive performance3. Further, Personalized Repetitive Transcranial Magnetic Stimulation (PrTMS) demonstrated increased efficacy in TMS treatments through utilizing quantitative electroencephalography (qEEG) and fine tuning the treatment to the individual. Yet, research examining the integration of PrTMS with assessments of sleep and cognition is scarce. Therefore, the main objective of this proposed study is to investigate the use of PrTMS, utilizing qEEG weekly for individualization, and the effects on sleep, cognitive performance, and overall wellness in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-42 years of age.

Exclusion Criteria:

* • Unable/unwilling to commit to participating in 1x per day treatments for 6 consecutive weeks

  * Outside of the age range of 18-42
  * Currently undergoing hormone therapy
  * History of blood clotting disorder
  * History of open skull traumatic brain injury
  * History of clinically significant seizure disorder
  * History of clinically significant manic episodes
  * Diagnosed with Diabetes Mellitus
  * Individuals with a clinically defined neurological disorder including, but not limited to:

    * Any condition likely to be associated with increased intracranial pressure
    * Space occupying brain lesion
    * History of cerebrovascular accident
    * Cerebral aneurysm
  * Has participated in any type of rTMS treatment within 3 months prior to the screening visit
  * Currently receiving antipsychotic or anticonvulsant medication treatment
  * Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed
  * Clinically significant medical illness, including any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning
  * History of psychosis
  * History of migraines
  * Current thoughts of suicidal ideation or self-harm
  * Substance use disorder within the past six months
  * Those pregnant or actively trying to become pregnant
  * Intake of one or a combination of the following drugs forms a 'Strong Potential Hazard' for application of rTMS due to their significant seizure threshold lowering potential:

    * Imipramine
    * Amitriptyline
    * Doxepine
    * Nortriptyline
    * Maprotiline
    * Chlorpromazine
    * Clozapine
    * Foscarnet
    * Ganciclovir
    * Ritonavir
    * Amphetamines
    * Cocaine (MDMA, ecstasy)
    * Phencyclidine (PCP, angel's dust)
    * Ketamine
    * Gamma-hydroxybutyrate (GHB)
    * Alcohol
    * Theophylline
    * Note: Being on one of these medications or substances would not automatically exclude a participant from study participation. The risk is dependent on the patient's past medical history, drug dose, speed of dose increase (or decrease), history of recent medication changes or duration of treatment, and combination with other CNS active drugs. Considering all the variables and keeping participant safety in mind, if a potential participant is on any of the above medication, the participant will be carefully evaluated and a justification for the decision to include them in the study will be documented by the medically responsible physician.
  * Recent withdrawal from one of the following drugs forms a 'Strong Relative Hazard' for application of rTMS due to the resulting significant seizure threshold lowering potential:

    * Alcohol
    * Barbiturates
    * Benzodiazepines
    * Meprobamate
    * Chloral hydrate

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Heart Rate as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Heart rate (beats per minute) will be quantified throughout the night via the OURA ring.
Change in Nocturnal Heart Rate Variability as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Heart rate variability (as measured by variance in time between heart beats) will be quantified throughout the night via the OURA ring.
Change in Sleep Latency as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Sleep onset latency will be quantified throughout the night via the OURA ring.
Change in Sleep Score as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Total sleep score will be quantified throughout the night via the OURA ring.
Change in Total Sleep Time as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Time of sleep will be quantified throughout the night via the OURA ring.
Change in Sleep Efficiency as measured by OURA Ring | Daily from baseline through study completion at 6 weeks
  Sleep efficiency will be quantified throughout the night via the OURA ring.
Change in Sleep Quality as measured via Questionnaire | Daily from baseline through study completion at 6 weeks
  A custom daily morning questionnaire will be used to record how a participant feels in regard to sleep restoration, recovery, and overall stress. This will be taken on the participants' smartphones within an hour of waking. Scores range from 3-10 with higher scores indicating poor sleep.
Change in Recovery as measured via Questionnaire | Daily from baseline through study completion at 6 weeks
  A custom daily morning questionnaire will be used to record how a participant feels in regard to sleep restoration, recovery, and overall stress. This will be taken on the participants' smartphones within an hour of waking. Scores range from 4-24 with higher scores indicating better recovery.
Change in Stress as measured via Questionnaire | Daily from baseline through study completion at 6 weeks
  A custom daily morning questionnaire will be used to record how a participant feels in regard to sleep restoration, recovery, and overall stress. This will be taken on the participants' smartphones within an hour of waking. Scores range from 4-24 with higher scores indicating more stress.
Change in Sustained Attention and Reaction Time | Daily from baseline through study completion at 6 weeks
  The Psychomotor Vigilance Task will be administered each morning within an hour of waking. This task will be completed on the participants' smartphone. Performance is calculated as 100% minus the number of lapses or false starts.
Change in Subjective Sleep Quality measured via Questionnaire | Weekly from baseline through study completion at 6 weeks.
  Participants will complete the Sleep Condition Indicator weekly. Scores range from 0-32. Higher scores indicate better sleep.
Change in Subjective Attention measured via Questionnaire | Intake (week 1), Mid-point (week 3) and exit (week 6)
  Participants will complete the Adult ADHD Self-Report Scale three different times. Scores are grouped by 0-16 = unlikely to have ADHD, 17-23 = likely to have ADHD, 24 or greater = highly likely to have ADHD.
Change in Subjective Anxiety measured via Questionnaire | Intake (week 1), Mid-point (week 3) and exit (week 6)
  Participants will complete the Hamilton Anxiety Rating Scale (HAM-A) three different times. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change in Subjective Depression measured via Hamilton Depression Rating Scale | Intake (week 1), Mid-point (week 3) and exit (week 6)
  Participants will complete the Hamilton Depression Rating Scale (HAM-D) three different times. The higher the score, the more severe the symptoms of depression. 10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Change in Subjective Depression measured via Patient Health Questionnaire | Intake (week 1), Mid-point (week 3) and exit (week 6)
  Participants will complete the Patient Health Questionnaire (PHQ-9) three different times. The higher the score, the more severe the symptoms of depression. Scores range from 5-9 = mild, 10-14 = moderate, 15-19 = moderate severe, 20-27 severe depression.
Change in Subjective Anxiety measured via Questionnaire | Weekly from baseline through study completion at 6 weeks
  Participants will complete the Generalzied Anxiety Disorder 7-item (GAD-7) scale weekly. Higher scores indicate anxious feelings. Scoring is grouped by 5-9 = mild, 10-14 = moderate, 15-21 = severe
Change in Mood as Indicated via Questionnaire | Daily from baseline through study completion at 6 weeks
  A custom daily morning questionnaire will be used to record how a participant feels in regard to mood and vigilance. Scores range from 8-100 with higher scores indicating better overall mood and vigilance.

CONTACTS AND LOCATIONS:
Locations (1):
- WVU Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States